CLINICAL TRIAL: NCT02152462
Title: Exergaming Intervention and Breast Cancer Biomarkers in Black Women
Acronym: POWER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Lucile Adams-Campbell, Principal Investigator, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00000116 Georgetown Lombard
Record Dates: First submitted 2014-03-31; First posted 2014-06-02 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer; Obesity
Keywords: exergaming; breast cancer; African American women; obesity
MeSH Terms: conditions — Breast Neoplasms; Obesity | interventions — Exergaming

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exergaming (Other): Exercise Intervention: Participants in the Wii Fit exergaming group will have a goal of 150 min/wk of moderate intensity exercise for the last 5 mo of the 6 mo intervention. Heart rate (HR) monitors will quantify exercise intensity. Participants will exercise at a HR equal to 45-65% of their VO2max. Participants will be instructed by the exercise physiologist on how to achieve the required HR. The training will consist of 3 days/wk of supervised Wii Fit physical activity. Exercise duration will increase gradually from 75 to 150 min/wk by wk 477. Thereafter, women will maintain >150 min/wk of moderate-intensity physical activity. Participants will complete daily exercise diaries recording the type and duration of physical activity, and HR.
  Interventions: Other: Exergaming
- Control (No Intervention): Control Group: After baseline testing the control group will be asked to maintain their current daily activities for the duration of the study. The control group will have the option to exercise at the Wii Fit stations following their completion of the study. They will receive the same measures as the exercise group.

INTERVENTIONS:
Other: Exergaming — The participants in the Wii Fit exergaming group will be encouraged to meet and then maintain a goal of 150 min/wk of moderate intensity exercise for 6 months. Goals per individual will be based on their baseline data. Exercise duration will increase gradually from 75 min/wk at week 1 to 150 min/wk by week 4. Thereafter, women will maintain >150 min/wk of moderate-intensity physical activity. The training will consist of 3 days/wk of supervised physical activity using Nintendo Wii Fit active videogames.
  Arms: Exergaming

SUMMARY:
Overview: This is a 6 month, two-arm randomized clinical trial using comparing exergaming to a control group. The investigators will randomize Black sedentary overweight/obese women to Wii Fit exercise (n=50) or the control arm (n=50). Women in the Wii Fit exercise group will come to the Georgetown community-based exercise facility 3 days/wk. The control group will be asked to maintain their current daily activities and not to exercise for the duration of the study. Based on the investigators previous findings that women who engage in 75-150 mins/wk of brisk walking had an 18% decreased risk of breast cancer, the investigators will target this level of activity in the investigators intervention arm. Also, this 150 min/week of physical activity meets the current recommendations of the American College of Sports Medicine (ACSM) and the US Department of Health and Human Services for healthy individuals and is in line with recommendation of the American Cancer Society (ACS) for cancer prevention.

DETAILED DESCRIPTION:
1. * Purpose of project (one or two sentences): To examine the feasibility and acceptability of an exergaming intervention in a community-based setting, and to explore the effects of exergaming on cardiovascular fitness, body mass index and percent body fat in Black women who are sedentary and overweight or obese.
2. * Study design (for example, hypothesis, research questions, standard and experimental procedures/drugs/devices or equipment, etc.):

Overview: This is a 6 month, two-arm randomized clinical trial using comparing exergaming to a control group. The investigators will randomize Black sedentary overweight/obese women to Wii Fit exercise (n=50) or the control arm (n=50). Women in the Wii Fit exercise group will come to the Georgetown community-based exercise facility 3 days/wk. The control group will be asked to maintain their current daily activities and not to exercise for the duration of the study. Based on the investigators previous findings that women who engage in 75-150 mins/wk of brisk walking had an 18% decreased risk of breast cancer, the investigators will target this level of activity in the investigators intervention arm. Also, this 150 min/week of physical activity meets the current recommendations of the American College of Sports Medicine (ACSM) and the US Department of Health and Human Services for healthy individuals and is in line with recommendation of the American Cancer Society (ACS) for cancer prevention.

Exercise Intervention: Participants in the Wii Fit exergaming group will have a goal of 150 min/wk of moderate intensity exercise for the last 5 mo of the 6 mo intervention. Heart rate (HR) monitors will quantify exercise intensity. Participants will exercise at a HR equal to 45-65% of their maximal oxygen consumption (VO2max). Given the expected VO2max values for this population, the investigators project that the Wii Fit videogames must elevate energy expenditure to 3-4 times resting metabolic rate to achieve the desired HR responses. As summarized above, previous studies have shown that such an elevation in energy expenditure can be expected from these activities. Wii Fit stations with a variety of active games will be available to participants at the Georgetown University Community Based Office. Participants will be instructed by the exercise physiologist on how to achieve the required HR. The training will consist of 3 days/wk of supervised Wii Fit physical activity. Exercise duration will increase gradually from 75 to 150 min/wk by wk 477. Thereafter, women will maintain >150 min/wk of moderate-intensity physical activity. Participants will complete daily exercise diaries recording the type and duration of physical activity, and HR.

Control Group: After baseline testing the control group will be asked to maintain their current daily activities for the duration of the study. The control group will have the option to exercise at the Wii Fit stations following their completion of the study. They will receive the same measures as the exercise group.

Diet: Participants in both groups will be instructed to maintain their diet constant throughout the study. Wii Fit intervention participants will be weighed at every session and those losing more weight than could be accounted for by their exercise will be counseled to return to their caloric intake at the start of the study.

* Rationale and justification for study (i.e. historical background, investigator's personal experience, pertinent medical literature, etc.): Several risk factors have been identified that increase breast cancer risk, some of which are non-modifiable factors (e.g., age, family history, and race) and some of which are modifiable (e.g., physical activity, body weight, dietary habits, and alcohol intake). However, only within the last 10 years have cancer organizations started to recommend physical activity as a preventive measure for breast cancer. The American Cancer Society (ACS) and the International Agency for Research on Cancer of the World Health Organization now both recommend regular physical activity as a strategy for women to reduce their risk of developing breast cancer. Specific recommendations for breast cancer prevention, which initially focused on diet, are now focused on maintaining a healthy weight throughout life by balancing caloric intake while increasing caloric expenditure via increased physical activity levels, and losing weight if overweight or obese. Obesity itself is a significant public health problem and is associated with increased postmenopausal breast cancer incidence and mortality. This research proposal will assess a novel method to improve physical activity in African American women, who are generally less physically active and more overweight and obese than women of most other racial and ethnic groups.

* Treatment Plan:

The participants in the Wii Fit exergaming group will be encouraged to meet and then maintain a goal of 150 min/wk of moderate intensity exercise for 6 months. Goals per individual will be based on their baseline data. Exercise duration will increase gradually from 75 min/wk at week 1 to 150 min/wk by week 4. Thereafter, women will maintain >150 min/wk of moderate-intensity physical activity. The training will consist of 3 days/wk of supervised physical activity using Nintendo Wii Fit active videogames.

Participants will exercise at a HR equal to 45-65% of their VO2max. Given the expected VO2max values for this population, the investigators project that the Wii Fit videogames will elevate energy expenditure to 3-4 times resting metabolic rate to achieve the desired HR responses. As summarized above, previous studies have shown that such an elevation in energy expenditure can be expected from these activities. Participants will be instructed to monitor their physical activity in order to assist with their perceived behavioral control and increase self-efficacy towards meeting their goals.

During aerobic exercise sessions, participants will wear Polar heart rate monitors to determine exercise intensity and will be given instruction by the exercise physiologist on how achieve the required HR. In addition, participants will complete daily exercise diaries to record the type and duration of physical activity, and exercise HR. Because many women may not have access to gym memberships or be able to afford expensive exercise equipment, the investigators address this environmental barrier by establishing Wii Fit stations with a variety of active games available to participants at the Community Based Office.

Exergames selected for use during the exercise sessions will be chosen based on energy expenditure data. Those active videogames that have been shown to achieve energy expenditure levels above those necessary to achieve 60% HRmax in the investigators specific study population will be selected. For example, active videogames tested in published studies, such as Wii Fit boxing and Dance Dance Revolution, have been found to achieve physical activity levels of moderate intensity (3.0-6.0 METs), which meet American College of Sports Medicine guidelines for health and fitness. Graves et al. (2008), for example found physical activity levels to reach 68% of maximal heart rate (HRmax) using the Wii Fit which also meets ACSM aerobic fitness recommendations (60% HRmax).

ELIGIBILITY:
Inclusion Criteria:

* Black women
* BMI ≥28 kg/m2 but ≤ 350 pounds of body weight
* Aged 40-59 years
* Sedentary (<60 min/wk exercise for past 6 months
* Never been diagnosed with cancer
* Ability to read and speak English and to provide meaningful consent
* No physical limitations preventing them from exercising
* Medical clearance by a health practitioner.

Exclusion Criteria:

* History of cancer
* Uncontrolled hypertension and medically treated diabetes
* Current enrollment in another physical activity and/or dietary study or a diet/weight loss program
* Pregnancy
* Inability to consent to study participation and complete assessments
* Telephone inaccessibility
* Physical limitations to exercise inability to commit to the intervention schedule

Ages: 40 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-12 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Biomarkers related to obesity and breast cancer risk | 6 months
  Outcomes for plasma leptin, adiponectin, Insulin-like growth factor 1 (IGF-1), Insulin-like growth factor-binding protein 3 (IGFBP3), C-reactive protein (CRP), Interleukin 6 (IL-6), insulin, c-peptide, and Hb-A1c levels at baseline and 24 weeks.

SECONDARY OUTCOMES:
Cardiovascular fitness (VO2 max) | 6 months
  Cardiovascular fitness is measured using metabolic cart at baseline, 12 weeks, and 24 weeks.
Reported stress levels | 6 months
  Reported stressed levels was assessed using the Perceived Stress Scale (PSS) at baseline, 12 weeks, and 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Lucile L Adams-Campbell, PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown Lombardi Office of Minority Health & Health Disparities Research, Washington D.C., District of Columbia, United States